CLINICAL TRIAL: NCT01134822
Title: Prospective Study of Fibrosis In the Lung Endpoints (PROFILE - Central England)
Acronym: PROFILE
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Medical Research Council (Other Government); GlaxoSmithKline (Industry); CRAFT Consortium (Unknown); McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: 09116
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2017-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; IPF; Lung Fibrosis; Biomarkers
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood(serum, plasma) & Lavage Fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Idiopathic pulmonary fibrosis (IPF)

SUMMARY:
The overall aim of this study is to develop a test that predicts the prognosis of IPF (Idiopathic Pulmonary Fibrosis) and which could be used to determine whether new treatments for IPF are likely to work.

DETAILED DESCRIPTION:
The overall objectives of this study are

* Discover and validate novel biomarkers and gene expression profiles for use in subsequent intervention studies in patients with IPF
* To prospectively validate a panel of previously published biomarkers in patients with well characterized idiopathic fibrosing lung disease
* Investigate genetic associations and epigenetic modifications which affect disease severity and progression
* Prospectively evaluate longitudinal disease behaviour in patients with IPF and NSIP with a view to developing composite clinical end-points for subsequent use in intervention studies in patients with IPF

Biomarkers that can be used for the following purposes will be identified:

* Identify patients (Diagnostic)(e.g. discriminate between health and disease)
* Correlate with disease severity (extent of disease, staging of disease)
* Predict clinical progression (Prognostic)(stable vs progressive disease)
* Track response to therapy (Therapeutic response)- Predict response to known efficacious treatments & Correlates with changes in clinical endpoints/mortality/quality of life
* Predict risk of exacerbations (could be used to prevent exacerbations or reduce their severity)
* Correlate with complications and/or comorbidities (e.g. biomarkers of Pulmonary Arterial Hypertension, Gastro Oesophageal Reflux in IPF, etc)

ELIGIBILITY:
Inclusion Criteria:

A diagnosis of IPF using the consensus criteria (32)and Non Specific Interstitial Pneumonia.

* Between the age group 18-85 years.
* Sub classified into Mild (TLCO>60), Moderate (TLCO 40-60), Severe (TLCO<40).
* People who volunteer to undergo a bronchoscopy for research

Exclusion Criteria:

* People who do not have IPF/NSIP (i.e. Hypersensitivity Pneumonitis, Sarcoidosis)
* People who cannot give informed consent.
* People who are being considered for bronchoscopy, any contra-indication to undergoing this procedure as set out in the British Thoracic Society guidelines (Thorax 2001; 56: suppl I: i1-i21). These will be part of the study but not undergo the Broncho Alveolar Lavage.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from IPF clinics
Sampling Method: Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2010-07; Primary Completion 2017-09-05 (Actual); Study Completion 2017-09-05 (Actual)

PRIMARY OUTCOMES:
Discover biomarkers in IPF | 36 months
  * Discover and validate novel biomarkers for use in subsequent intervention studies in patients with IPF
  * To prospectively validate a panel of previously published biomarkers in patients with well characterized idiopathic fibrosing lung disease
  * Investigate genetic associations and epigenetic modifications which affect disease severity and progression

SECONDARY OUTCOMES:
Survival from Pulmonary fibrosis. | 10 years
  All patients will be tagged at the central NHS registry in order to provide mortality data. For this reason we will need to keep our datasets active for up to 10 years to allow a complete mortality analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Gisli Jenkins, Dr, Study Director — University of Nottingham; Robert Berg, Dr, Principal Investigator — University Hospitals of Derby and Burton NHS Foundation Trust; Sanjay Agarwal, Dr, Principal Investigator — University Hospitals, Leicester; Moira White, Dr, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust; Khaled Amsha, Dr, Principal Investigator — Sherwood Forest Hospitals NHS Trust; David Thickett, Dr, Principal Investigator — University Hospital Birmingham NHS Foundation Trust; Uttam Nanda, Dr, Principal Investigator — Burton Hospitals NHS Foundation Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allen RJ, Stockwell A, Oldham JM, Guillen-Guio B, Schwartz DA, Maher TM, Flores C, Noth I, Yaspan BL, Jenkins RG, Wain LV; International IPF Genetics Consortium. Genome-wide association study across five cohorts identifies five novel loci associated with idiopathic pulmonary fibrosis. Thorax. 2022 Aug;77(8):829-833. doi: 10.1136/thoraxjnl-2021-218577. Epub 2022 Jun 10. PMID 35688625
- [Derived] Clynick B, Corte TJ, Jo HE, Stewart I, Glaspole IN, Grainge C, Maher TM, Navaratnam V, Hubbard R, Hopkins PMA, Reynolds PN, Chapman S, Zappala C, Keir GJ, Cooper WA, Mahar AM, Ellis S, Goh NS, De Jong E, Cha L, Tan DBA, Leigh L, Oldmeadow C, Walters EH, Jenkins RG, Moodley Y. Biomarker signatures for progressive idiopathic pulmonary fibrosis. Eur Respir J. 2022 Mar 31;59(3):2101181. doi: 10.1183/13993003.01181-2021. Print 2022 Mar. PMID 34675050
- [Derived] Maher TM, Oballa E, Simpson JK, Porte J, Habgood A, Fahy WA, Flynn A, Molyneaux PL, Braybrooke R, Divyateja H, Parfrey H, Rassl D, Russell AM, Saini G, Renzoni EA, Duggan AM, Hubbard R, Wells AU, Lukey PT, Marshall RP, Jenkins RG. An epithelial biomarker signature for idiopathic pulmonary fibrosis: an analysis from the multicentre PROFILE cohort study. Lancet Respir Med. 2017 Dec;5(12):946-955. doi: 10.1016/S2213-2600(17)30430-7. Epub 2017 Nov 14. PMID 29150411
- [Derived] Jenkins RG, Simpson JK, Saini G, Bentley JH, Russell AM, Braybrooke R, Molyneaux PL, McKeever TM, Wells AU, Flynn A, Hubbard RB, Leeming DJ, Marshall RP, Karsdal MA, Lukey PT, Maher TM. Longitudinal change in collagen degradation biomarkers in idiopathic pulmonary fibrosis: an analysis from the prospective, multicentre PROFILE study. Lancet Respir Med. 2015 Jun;3(6):462-72. doi: 10.1016/S2213-2600(15)00048-X. Epub 2015 Mar 12. PMID 25770676